CLINICAL TRIAL: NCT06498505
Title: HighCycle: Effect of Acetazolamide on Pulmonary Artery Pressure in Women Compared to Men. A Randomized, Placebo-Controlled, Double-Blind Parallel Trial.
Brief Title: HighCycle: Effect of Acetazolamide on Pulmonary Artery Pressure in Women Compared to Men
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government); University Hospital Heidelberg (Other); Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HighCycle_PAP
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: High Altitude
Keywords: Women; Hypoxia; Prevention; Acetazolamide; Echocardiography
MeSH Terms: conditions — Altitude Sickness; Hypoxia | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- WOMEN - ACETAZOLAMIDE oral capsule (Active Comparator): Acetazolamide 250 mg/day (capsules @125 mg; 1 in the morning, 1 in the evening), orally. Medication starts 24 hours before ascent to 3600 m until the morning after the second night at 3600 m
  Interventions: Drug: Acetazolamide
- MEN - ACETAZOLAMIDE oral capsule (Active Comparator): Acetazolamide 250 mg/day (capsules @125 mg; 1 in the morning, 1 in the evening), orally. Medication starts 24 hours before ascent to 3600 m until the morning after the second night at 3600 m
  Interventions: Drug: Acetazolamide
- WOMEN - PLACEBO oral capsule (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules; 1 in the morning, 1 in the evening), orally. Medication starts 24 hours before ascent to 3600 m until the morning after the second night at 3600 m.
  Interventions: Drug: Placebo
- MEN - PLACEBO oral capsule (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules; 1 in the morning, 1 in the evening), orally. Medication starts 24 hours before ascent to 3600 m until the morning after the second night at 3600 m.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Administration of 1x125mg acetazolamide in the morning, 1x125mg in the evening, starting 24 hours before departure to 3600 m.
  Arms: MEN - ACETAZOLAMIDE oral capsule; WOMEN - ACETAZOLAMIDE oral capsule
Drug: Placebo — Administration of equally looking placebo capsules in the morning and in the evening, starting 24 hours before departure to 3600 m.
  Arms: MEN - PLACEBO oral capsule; WOMEN - PLACEBO oral capsule

SUMMARY:
Randomized clinical trial evaluating the effect of acetazolamide on pulmonary artery pressure in women compared to men travelling to 3600 m.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking men and women, age 18-44 years, without any diseases and need of regular medication (including oral contraceptives).
* BMI >18 kg/m2 and <30 kg/m2
* Born, raised and currently living at altitudes <1000 m
* Written informed consent
* Premenopausal women with an eumenorrheic cycle

Exclusion Criteria:

* Other types of contraceptvies (hormonal intrauterine device, vaginal ring, subcutaneous injections or implants, among others)
* Pregnancy or nursing
* Anaemic (haemoglobin concentration <10g/dl)
* Any altitude trip <4 weks before the study
* Allergy to acetazolamide and other sulfonamides

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary artery Pressure (PAP) | Day 2 at 760 m and Day 2 at 3600 m
  Sex-related difference in the altitude-induced change in RV/RA in mmHg assessed by echocardiography between acetazolamide and placebo group.

SECONDARY OUTCOMES:
Lung comets | Day 2 at 760 m and Day 2 at 3600 m
  Sex-related difference in the altitude-induced change in ultrasound lung comets assessed by echocardiography between acetazolamide and placebo group.
Parameters of right heart function | Day 2 at 760 m and Day 2 at 3600 m
  Sex-related difference in the altitude-induced change in parameters of right heart function assessed by echocardiography between acetazolamide and placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof. Dr., Study Chair — University of Zurich; Talant Sooronbaev, Prof. Dr., Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center for Cardiology and Internal Medicine, Bishkek, Gorod Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided